CLINICAL TRIAL: NCT00487981
Title: Precision Spinal Cord Stimulation for Painful Diabetic Neuropathy
Brief Title: Spinal Cord Stimulation for Painful Diabetic Neuropathy
Acronym: DPN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient Data Collected
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS0206
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-02

CONDITIONS: Diabetic Neuropathy; Pain; Peripheral Neuropathy
Keywords: Pain; Implantable stimulation device; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spinal Cord Stimulation Group (Other): Spinal Cord Stimulation (SCS) Treatment Group
  Interventions: Device: Precision Spinal Cord Stimulation

INTERVENTIONS:
Device: Precision Spinal Cord Stimulation — Stimulation on throughout the study once device is implanted
  Other Names: Precision Spinal Cord Stimulation System

SUMMARY:
The purpose of this study is to evaluate Spinal Cord Stimulation (SCS) therapy in individuals who suffer from painful diabetic peripheral neuropathy. Patients invited to participate in this study will be eligible for SCS therapy, and will have already selected therapy with the Advanced Bionics Precision system independent of possible inclusion in this study. The device, accessories, and procedures associated with device placement and the indications for use are all consistent with the current and approved product labeling.

DETAILED DESCRIPTION:
The management of neuropathic pain is often difficult, and the available treatment options rarely provide complete relief. Although prevention by means of glycemic control is the first priority, up to 20% of patients will develop Diabetic Peripheral Neuropathy (DPN) and require active drug therapy. Select anti-depressants, anti-epileptics, and opioids have generally been the first-line pharmacologic treatments for neuropathic pain. Topical creams have been used to achieve local control. Nonconventional therapies have included acupuncture and magnet therapy. However, all of these treatments have limited utility because of marginal efficacy. Various forms of electric stimulation have been shown to improve the symptoms of DPN. Advances in spinal cord stimulation technology have encouraged broader use of this treatment modality in the management of chronic painful DPN.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic neuropathic pain in at least one limb with a score of at least 3 using the Michigan Neuropathy Screening Instrument (MNSI) secondary to Type 1 or Type 2 diabetes
* Have chronic neuropathic pain for at least 12 months
* Be 18 years of age or older
* Be refractory to pain medication including gabapentin or the use of pain medication is contraindicated or not tolerated because of side effects or other medical condition
* Be an appropriate candidate for SCS therapy and have already decided to use the Precision system
* Be willing and able to comply with all study related procedures and visits
* Be capable of reading and understanding patient information materials and giving written informed consent

Exclusion Criteria:

* Are a smoker
* Have any other chronic pain condition likely to confound evaluation of study endpoints
* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints such as peripheral vascular disease or neurological disorders unrelated to diabetic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis McDonnell, MD, Principal Investigator — Deaconess Hospital
Locations (1):
- Deaconess Pain Management Center, Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation (SCS) Group: Spinal Cord Stimulation (SCS) Treatment Group
Period: Overall Study
Arm/Group | Spinal Cord Stimulation (SCS) Group
Started | 1
Completed | 0
Not Completed | 1
Not completed — Hypothyroidism diagnosis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Cord Stimulation (SCS) Group
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating at 6 Months Post Activation Compared to Baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percent reduction
Arm/Group | Spinal Cord Stimulation (SCS) Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Spinal Cord Stimulation (SCS) Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
One subject enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less